CLINICAL TRIAL: NCT05831280
Title: The Effect of Laughter Yoga on the Stress Levels of Infertility Women: A Randomized Controlled Trial
Brief Title: The Effect of Laughter Yoga on the Stress Levels of Infertility Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aslı SİS ÇELİK, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: aslı14
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Laughter Yoga
Keywords: Laughter Yoga; Infertility; Stress; Nurse
MeSH Terms: conditions — Infertility | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The women in the experimental and control groups did not know which group they were in. Data were collected online due to the pandemic. Therefore, the researchers and the people who would conduct the analyzes did not know the women in the experimental and control groups. The women used a nickname to fill in the questions on the measurement tools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimantal Group (Experimental): In the study, 8 sessions of laughter yoga will be applied to the women in the experimental group twice a week for 4 weeks.
  Interventions: Behavioral: Laughter Yoga
- Control Group (No Intervention): no intervention will be applied to the control group

INTERVENTIONS:
Behavioral: Laughter Yoga — * Warm-up exercises (5 minutes),
  * Deep breathing exercises (5 minutes),
  * Childlike playfulness (5 minutes),
  * Laughter exercises (15 minutes).
  Arms: Experimantal Group

SUMMARY:
This research is a randomized controlled study to evaluate the effect of Laughter yoga on the stress levels of infertility women. Randomization was provided in the sample included in the study, and it was divided into experimental and control groups. At the beginning of the study, the Infertility Stress Scale was applied to women in both groups to determine their stress levels. Afterwards, 8 sessions of laughter yoga were applied to the experimental group for 4 weeks. No application was made to the control group. After 4 weeks, the Infertility Stress Scale was administered to the women in both groups to re-determine their stress levels.

DETAILED DESCRIPTION:
This research is a randomized controlled study to evaluate the effect of Laughter yoga on the stress levels of infertility women. At the beginning of the study, necessary ethics committee permission and institutional permissions were obtained. Both of the researchers have a certificate of leadership in laughter yoga. As a result of the power analysis, it was determined that 80 women should be included in the study. Considering that there may be losses, it was decided to include 90 women in the study. By providing randomization, 90 women who met the sampling criteria and volunteered to participate in the study were divided into two groups as 45 experimental and 45 control. At the beginning of the study, the Infertility stress scale was applied to women in both groups to determine their stress levels. Afterwards, 8 sessions of laughter yoga were applied to the experimental group for 4 weeks, two sessions a week. No application was made to the control group. After 4 weeks, the Infertility stress scale was administered to the women in both groups to re-determine their stress levels.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 19-45
* have been diagnosed with infertility
* At least primary school graduate
* Not having a diagnosed psychiatric disease
* Will not have an ovulation pick up process, Intrauterine insemination and Embryo transfer procedure in the next 1 month

Exclusion Criteria:

* Have ovulation pick up process in the last 1 month
* undergoing Intrauterine insemination in the last 1 month
* undergoing an Embryo transfer in the last 1 month
* Not regularly attending laughter yoga sessions (for the experimental group)
* Applying another alternative method to reduce stress during the research process

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Stress levels of women | 1 month
  The difference between the infertility stress scale pretest and posttest mean scores of women in both groups. Higher scores indicate increased stress.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı SİS ÇELİK, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Yakutiye, Turkey (Türkiye)